CLINICAL TRIAL: NCT00739960
Title: Sarcoidosis, Trial of Abatacept in Refractory Disease (STAR). A Prospective Open-Label Trial of Abatacept in Progressive Sarcoidosis
Brief Title: Safety Study of Abatacept to Treat Refractory Sarcoidosis
Acronym: STAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding has been pulled
Sponsor: University of Chicago (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: University of Chicago #15630B
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abatacept (Other)
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — 10mg/kg IV (infusion directly into the vein of the arm) Day 1, week 2, week 4 and then every 4 week for 44 weeks.
  Other Names: Orencia

SUMMARY:
The purpose of this study is to determine how safe and effective Abatacept is in treating patients who have progressive pulmonary sarcoidosis.

ELIGIBILITY:
Primary Inclusion Criteria:

* Diagnosis of sarcoidosis for at least 1 year with lung disease
* Active disease despite current treatment
* On a stable dose of sarcoidosis treatment with oral steroids, methotrexate, or hydroxychloroquine, for at least 90 days

Primary Exclusion Criteria:

* Previous treatment with Abatacept
* Currently receiving or received within the last 60 days the following: TNFα-inhibitors (infliximab, etanercept, adalimumab)
* Currently receiving or received within the last 30 days the following: cyclosporine, tacrolimus or leflunomide
* Previous treatment of IVIg within the last 6 months
* History of chronic infection that has been active within last 60 days, or herpes zoster within last 6 months, or any infection requiring hospitalization or intravenous medication within last 60 days or oral medication within the last 2 weeks
* History of congestive heart failure
* HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadera J Sweiss, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abatacept
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Open Label: Open label for Abatacept
Arm/Group | Open Label
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety of Abatacept in Progressive Pulmonary Sarcoidosis.
Description: Adverse events that are considered by the investigator to be reasonably or probably related to Abatacept.
Time Frame: 24 weeks and 52 weeks
Population: Since this study was designed to be a safety study, we chose safety as the primary outcome. Any change of symptoms from baseline was considered possibly related to the study drug, although unlikely. The study was discontinued due to funding withdrawal caused by the principal investigator switching institutions.
Measure: Number; unit: participant adverse events
Arm/Group | Abatacept
Number analyzed (Participants) | 1
participant adverse events | 1

2. Secondary Outcome: Change From Baseline in 6-minute Walk Distance.
Time Frame: 24 weeks and 52 weeks
Population: Data was not collected for this Outcome Measure.
Arm/Group | Abatacept
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 weeks.
Description: No serious adverse events were reported.
Arm/Group | Abatacept
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=1)
Worsening shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — The patient had advanced fibrotic pulmonary sarcoidosis. It was unclear whether the worsening shortness of breath was due to the disease or to the study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No